CLINICAL TRIAL: NCT00003187
Title: The Unrelated Donor Marrow Transplantation Trial
Brief Title: Bone Marrow Transplantation in Treating Patients With Leukemia, Myelodysplasia, or Lymphoblastic Lymphoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Saul Yanovich, MD, Virginia Commonwealth University/Massey Cancer Center
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066016; P30CA016059 (NIH); MCV-CCHR-9504-2X; DUMC-75951; NCI-G98-1388
Record Dates: First submitted 2000-05-02; First posted 2004-05-24 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes
Keywords: recurrent childhood acute lymphoblastic leukemia; stage IV childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; untreated childhood acute lymphoblastic leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; acute undifferentiated leukemia; stage IV adult lymphoblastic lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Leukemia, Biphenotypic, Acute | interventions — Filgrastim; Cyclophosphamide; Cyclosporine; Cytarabine; Methotrexate; Methylprednisolone; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: cyclosporine
Drug: cytarabine
Drug: methotrexate
Drug: methylprednisolone
Procedure: allogeneic bone marrow transplantation
Procedure: in vitro-treated bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Bone marrow transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy used to kill cancer cells. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Eliminating the T cells from the donor cells before transplanting them may prevent this from happening.

PURPOSE: Randomized phase II/III trial to compare the effectiveness of conventional bone marrow transplantation with T cell-depleted bone marrow transplantation in treating patients who have leukemia, myelodysplasia, or lymphoblastic lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the disease free survival of patients with leukemia, myelodysplasia, or lymphoblastic lymphoma after treatment with conventional (non-T cell depleted) or T cell depleted unrelated donor bone marrow transplantation. II. Compare the incidence of primary and secondary graft failure, acute and chronic graft-vs-host disease, complications (infection, veno-occlusive disease, interstitial pneumonitis), and relapse in these patients after these treatments. III. Compare the incidence of other malignancies, lymphoproliferative disorders, and post-transplant myelodysplasia in these patients after these treatments.

OUTLINE: This is a randomized, multicenter study. Patients will be stratified according to institution. Patients are assigned to one of two treatment arms, one with conventional bone marrow transplantation (arm I) and one with T cell depletion of the bone marrow (arm II). Arm I: Patients receive cyclophosphamide on days -6 and -5. Total body irradiation (TBI) is administered on days -4 to 0, although this order may be reversed. Males with ALL receive a testicular boost of radiation therapy. Bone marrow is infused on day 0. Patients receive cyclosporine beginning on day -1 and methotrexate IV on days 1, 3, 6, and 11. Arm II: T cell depletion is conducted by 2 different methods, according to the institution, and treatment varies depending on the method used. Method I is by T10B9 depletion and Method II is by counterflow elutriation depletion. Method I: Depending on the institution, some patients receive TBI on days -9 to -7 (before chemotherapy) (Course I) and some receive TBI on days -3 to -1 (after chemotherapy) (Course II). Course I also includes cytarabine IV on days -5 to -3, cyclophosphamide IV on days -2 and -1, and methylprednisolone IV on days -2 to 0 and 5-18. Bone marrow infusion is administered on day 0. Cyclosporine begins on day -1. Course II includes cytarabine IV on days -7 to -4 and cyclophosphamide on days -6 to -5. Methylprednisolone IV is administered on days -2 to 0 and 5-18. Bone marrow infusion is administered on day 0. Cyclosporine begins on day 0. Method II: Preparative therapy varies according to the disease category. Acute lymphoblastic leukemia: Patients undergo TBI on days -7 to -4. Males receive testicular boost on day -7, and all receive electron boost to anterior and posterior chest wall on days -5 and -4. Cyclophosphamide IV is administered on days -3 and -2. Bone marrow infusion is administered on day 0. Acute nonlymphocytic leukemia, chronic myelogenous leukemia, and myelodysplastic syndrome: Patients receive cyclophosphamide IV on days -7 and -6, followed by TBI on days -4 to -1. Bone marrow infusion is administered on day 0. Patients receive methylprednisolone IV every 12 hr on days -2,-1, and 5-19. Cyclosporine is administered from day -3 to day 180. All patients on both arms receive filgrastim (granulocyte colony-stimulating factor; G-CSF) beginning on day 7 post-transplant. Patients are followed weekly for the first 14 weeks, at day 100, every 6 months for 2 years, then annually thereafter.

PROJECTED ACCRUAL: A total of 560 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Pathologically confirmed acute myeloid leukemia Not in first complete remission with translocations t(8;21) unless failed first line induction therapy Not in first complete remission with translocations t(15;17) or 16q abnormality unless: Failed first line induction therapy OR Molecular evidence of disease Pathologically confirmed acute lymphoblastic lymphoma (ALL) Not in first complete remission OR High risk ALL in first complete remission defined as: Hypodiploidy OR Pseudodiploidy with translocations t(9,22), t(4;11), or t(8;14) OR Elevated WBC at presentation Greater than 100,000/mm3 if 6-12 months old Greater than 50,000/mm3 if 10-20 years old Greater than 20,000/mm3 if 21 or over OR Failed to achieve complete remission after 4 weeks of induction therapy Pathologically confirmed chronic myelogenous leukemia (CML) not in blast crisis Pathologically confirmed undifferentiated leukemia or biphenotypic leukemia Pathologically confirmed juvenile CML with or without either 7q- or infantile monosomy 7 Leukocytosis with absolute monocytosis greater than 450 microliters AND Immature myeloid cells in peripheral blood circulation Less than 25% marrow blasts Myelodysplastic syndromes: Refractory anemia (RA) RA with ringed sideroblasts RA with excess blasts (RAEB) RAEB in transformation Chronic myelomonocytic leukemia Pathologically confirmed stage IV lymphoblastic lymphoma No active CNS or skin leukemic involvement No consenting suitably HLA-matched related donor available Consenting unrelated donor available

PATIENT CHARACTERISTICS: Age: 55 and under Performance status: Karnofsky 70-100% OR Lansky 60-100% Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Bilirubin less than 2.5 mg/dL SGOT less than 3 times upper limit of normal Renal: Creatinine within normal range OR Creatinine clearance greater than 60 mL/min Cardiovascular: Asymptomatic OR Left ventricular ejection fraction at rest greater than 40% and improves with exercise Pulmonary: Asymptomatic OR DLCO greater than 45% Other: Not pregnant or lactating HIV negative No uncontrolled viral, bacterial, or fungal infection

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior autologous or allogeneic bone marrow transplant Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: No concurrent mediastinal radiation No prior radiation therapy that would preclude total body irradiation Surgery: Not specified

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 1995-05; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ann Jensen, PhD, Study Chair — National Heart, Lung, and Blood Institute (NHLBI)
Locations (13):
- United States (13):
  - Stanford University Medical Center, Stanford, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - University of South Carolina School of Medicine, Columbia, South Carolina
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Massey Cancer Center, Richmond, Virginia
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Lehtoranta L, Hibberd AA, Yeung N, Laitila A, Maukonen J, Ouwehand AC. Characterization of vaginal fungal communities in healthy women and women with bacterial vaginosis (BV); a pilot study. Microb Pathog. 2021 Dec;161(Pt A):105055. doi: 10.1016/j.micpath.2021.105055. Epub 2021 Jun 17. PMID 34146644